CLINICAL TRIAL: NCT03294057
Title: The Effectiveness of Collaborative Care With Smart Health Management Program for Patients With Chronic Illness: Randomized Controlled Trial
Brief Title: Collaborative Care With Smart Health Management Program for Patients With Chronic Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korea Health Industry Development Institute (Other Government); National Evidence-Based Healthcare Collaborating Agency (Other Government); National Institute of Health, Korea (Other Government); National Clinical Research Coordination Center, Seoul, Korea (Other Government); Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Young Ho Yun, Principal Investigator, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HI16C0455-2
Record Dates: First submitted 2017-09-19; First posted 2017-09-26 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Osteoporosis; Chronic Respiratory Disease; Arthritis; Osteopenia
Keywords: Self-Management IT Program
MeSH Terms: conditions — Osteoporosis; Arthritis; Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ICT programs + Tele-coaching programs (Experimental): ICT programs that include health information learning by disease and self-management based on Smart Management Strategy for Health (SMASH) are provided. And a trained nurse provides tele-coaching programs to subjects. After that, subjects will conduct self-management health care and tele-coaching programs for 12 weeks. After 3 months, they finish self-management ICT + coaching programs, and then they fill out the questionnaire.
  Interventions: Behavioral: Tele-coaching programs; Behavioral: ICT programs
- ICT programs (Experimental): ICT programs that include health information learning by disease and self-management based on Smart Management Strategy for Health (SMASH) are provided. After that, subjects will conduct self-management health care for 12 weeks. After 3 months, they finish self-management ICT programs, and then they fill out the questionnaire.
  Interventions: Behavioral: ICT programs
- A book about chronic disease (Active Comparator): Subjects in the group get a book about chronic disease for patients. After 3 months, they finish reading the materials, they fill out the questionnaire.
  Interventions: Behavioral: A book about chronic disease

INTERVENTIONS:
Behavioral: Tele-coaching programs — Tele-coaching program conducted 12 times (one time for one week), and more than 20 minutes each by a trained nurse. Coaching content specifically, 1) evaluation, 2) facing and accepting the health crisis, 3) setting up new goals, 4) making decisions and plans, and 5) practice.
  Arms: ICT programs + Tele-coaching programs
Behavioral: ICT programs — ICT programs that include health information learning by disease and self-management based on Smart Management Strategy for Health (SMASH)
  Arms: ICT programs; ICT programs + Tele-coaching programs
Behavioral: A book about chronic disease — A Take-home book about chronic disease are provided for self-education
  Arms: A book about chronic disease

SUMMARY:
This study verifies efficacy of collaborative care with Smart Health Management Program developed for patients with chronic illness. The aim of the study is to observe the changes in clinical indicators, quality of life and health related behaviors when providing self-management programs with ICT for chronic disease patients.

DETAILED DESCRIPTION:
This study is to demonstrate that chronic disease patients receiving collaborative care with ICT-based self-management and educational program can improve clinical outcomes and overall health status, including quality of life and health habits.

In addition to the economic burden, people with chronic disease experience various psychosocial crises such as anxiety and depression, which causes the deterioration of overall quality of life and increases social burden. The collaborative care management based Chronic Care Model (CCM) have provided coaching by a medically supervised nurse, working with each patient's physician. However, standard CCM have limitations in that they do not provide self-management strategies of the patient in detail. Therefore, to improve the effectiveness of the CCM model, it is required to propose a new approach to the utilization of IT-based self-management program that is currently being developed to increase accessibility and efficiency of health care service.

Primary outcomes of this study are as follow: Improvement of depression in patients with osteoporosis, chronic respiratory disease and chronic arthritis.

Participants in this study will respond a baseline questionnaire about depressive mood, health habits, health behavior patterns and quality of life, diet, exercise, etc. After that, participants will be allocated equally into three groups - the intervention group 1, intervention group 2 and the control group. The intervention group 1 will receive S Healthing and a tele- coaching program conducted 12 times (one time for one week), and more than 20 minutes each by a trained nurse. The intervention group 2 will receive S Healthing while the control group will receive basic educational material on the disease. Coaching content consists specifically of: 1) evaluation, 2) facing and accepting the health crisis, 3) setting up new goals, 4) making decisions and plans, and 5) practice. "S Healthing" is based ICT- program and includes educational contents and self-management program based on Smart Management Strategy for Health (SMASH). The intervention group 1, 2 will conduct self-management for 3 months through smart phone application and web program. Participants will receive a questionnaire about the quality of life and health habits with the clinical examination 3 months after baseline survey was conducted. The result from two questionnaires (baseline, 3 months post-intervention) and clinical outcome of baseline and 3 months will be compiled and be compared with others.

ELIGIBILITY:
Inclusion Criteria:

* Subject 19 years old and more
* Subject who understands the purpose of the study and signs with informed consent form
* Subject with chronic disease (osteoporosis, chronic pulmonary disease, chronic arthritis)
* Subject with METs less than 12.5 hours per week
* Subjects who use smart phones and PCs (those who can use ICT-based health care programs)

Exclusion Criteria:

* Inability to speak, understand, or write Korean
* Inability to understand the contents of the provided materials due to poor eyesight and hearing
* Medical conditions that would limit adherence to participation of the clinical trial (as confirmed by their referring physician; e.g. dyspnea, severe depression and other mental disorders)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Depression | Baseline, 3 months post-intervention
  Improvement of depression (PHQ-9)

SECONDARY OUTCOMES:
Health behavior patterns | Baseline, 3 months post-intervention
  We identify health habits by dividing into five steps according to the TTM stage. We evaluate Increase in maintenance rate of health behavior patterns.
Health Management Strategies | Baseline, 3 months post-intervention
  Improvement of Health Management Strategies by SAT (We use Smart Management Strategy for Health Assessment Tool (SAT) to assess their self-management (SM) strategies of health by themselves).
Quality of life (Mcgill QoL) | Baseline, 3 months post-intervention
  Improvement of quality of life (Mcgill QoL)
Quality of life (EuroQoL) | Baseline, 3 months post-intervention
  Improvement of quality of life (EuroQoL)
Quality of life (SF-12) | Baseline, 3 months post-intervention
  Improvement of quality of life (SF-12)
Physical activity | Baseline, 3 months post-intervention
  Changes in exercise (Godin's Leisure Time Exercise Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Young Ho Yun, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kang E, Park SM, Lee K, Lee EB, Yim JJ, Lee J, Kim S, Rhee YE, Yun YH. Efficacy of Health Coaching and an Electronic Health Management Program: Randomized Controlled Trial. J Gen Intern Med. 2021 Sep;36(9):2692-2699. doi: 10.1007/s11606-021-06671-2. Epub 2021 Mar 5. PMID 33674921